CLINICAL TRIAL: NCT04801862
Title: Clinical, Microbiological and Genetic Factors Associated With Recurrence of Clostridioides Difficile Infection and Development of a Predictive Tool for Recurrence
Brief Title: Natural History of Clostridioides Difficile Infection
Status: Recruiting | Type: Observational
Sponsor: Hospital Universitario de Valme (Other)
Responsible Party: Principal Investigator, Nicolás Merchante, Coordinator of the UCEIM-HUV Research Group, Hospital Universitario de Valme
Other Study IDs: PI20/01450
Record Dates: First submitted 2021-03-12; First posted 2021-03-17 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Clostridium Difficile Infection; Health Care Associated Infection; Nosocomial Infection
Keywords: Clostridioides difficile; Clostridium difficile; Nosocomial diarrhea; Health care associated infection; Nosocomial infection; Antimicrobial stewardship
MeSH Terms: conditions — Clostridium Infections; Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — Blood sample for genetic studies and stool samples for microbiological studies
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed of C.difficile infection: Open cohort of consecutive patients diagnosed of Clostridioides difficile infection

SUMMARY:
Aim: To investigate if host factors, such as composition and diversity of intestinal microbiota and/or genetic determinants, are associated with a higher risk of recurrence of Clostridioides difficile infection (CDI). To generate a predictive tool based on epidemiological, clinical, genetic and microbiologic variables aimed to identify patients at a higher risk of CDI recurrence in a context of optimized ICD management. Design: Multicenter prospective cohort study. Patients: Older than 18 years patients with CDI diagnosis, made by IDSA criteria, in the participant centers.

Follow-up: A stewarship program aimed to improve CDI management, including early detection of CDI recurrence, will be implemented in the participant centers. Blood samples for genetic testing and stool samples for intestinal microbiome studies will be collected.

Variables and data analysis: The primary outcome variable will be the emergence of CDI recurrence. Potential independent predictors of recurrence, including genetic and microbiological factors, will be assessed. A predictive tool based on independent predictors of recurrence will be built in a development subpopulation. The performance of the model will be assessed by ROC curves, and sensititvity, especificity, as well as negative and positive predictive values will be calculated, both in the development subpopulation and in a validation subset.

ELIGIBILITY:
Inclusion Criteria:

* Age older than 18 years
* New episode of Clostridioides difficile infection, based on IDSA criteria.

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed of Clostridoides difficile infection
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
CDI recurrence | First 8 weeks after end of therapy
  Clostridioides difficile recurrence
CDI reinfection | Between 8 weeks after end of therapy and before 24 weeks
  New episode of Clostridioides difficile infection

SECONDARY OUTCOMES:
Readmission due to CDI infection | During 24 weeks after the end of therapy
  New hospitalization related to new Clostridioides difficile infection episode

CONTACTS AND LOCATIONS:
Locations (15):
- Spain (15):
  - Hospital Vega Baja, Orihuela, Alicante
  - Hospital Marina Baixa, Villajoyosa, Alicante
  - Hospital Universitario de Puerto Real, Puerto Real, Cadiz
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario San Juan, Alicante
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Universitario San Cecilio, Granada
  - Hospital Juan Ramón Jiménez, Huelva
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario de Valme, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Consorcio Hospital General de Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Politécnico Universitario La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Merchante N, Herrero R, Valverde-Fredet MD, Rodriguez-Fernandez M, Pinagorte H, Martinez-Marcos FJ, Gil-Anguita C, Garcia-Lopez M, Tasias Pitarch M, Abril Lopez De Medrano V, Navarrete Lorite MN, Gomez-Ayerbe C, Leon E, Gonzalez-De La Aleja P, Ruiz Castillo A, Aller AI, Rodriguez JC, Ternero Fonseca J, Corzo JE, Naranjo Perez A, Trigo-Rodriguez M, Merino E. Role of previous systemic antibiotic therapy on the probability of recurrence after an initial episode of Clostridioides difficile infection treated with vancomycin. JAC Antimicrob Resist. 2023 Mar 23;5(2):dlad033. doi: 10.1093/jacamr/dlad033. eCollection 2023 Apr. PMID 36968953
- [Background] Merchante N, Chico P, Marquez-Saavedra E, Riera G, Herrero R, Gonzalez-de-la-Aleja P, Aller AI, Rodriguez JC, Rodriguez-Fernandez M, Ramos JM, Trigo-Rodriguez M, Merino E. Impact of COVID19 pandemic on the incidence of health-care associated Clostridioides difficile infection. Anaerobe. 2022 Jun;75:102579. doi: 10.1016/j.anaerobe.2022.102579. Epub 2022 Apr 30. PMID 35500744
- [Derived] Rodriguez-Fernandez M, Herrero R, Gonzalez-De-La-Aleja P, Valverde-Fredet MD, Ventero MP, Trigo-Rodriguez M, Giner L, Aller-Garcia AI, Pinargote-Celorio H, Espindola-Gomez R, Parra M, Martinez Perez-Crespo P, Ramos-Rincon JM, Fernandez-Pevida A, Lanz-Garcia J, Leon E, Valiente-De-Santis L, Corzo JE, Rodriguez JC, Merino E, Merchante N. Clinical Impact of Implementing a Specific Clinical Pathway for the Management of Clostridioides difficile Infection. Infect Dis Ther. 2025 Nov 7. doi: 10.1007/s40121-025-01261-9. Online ahead of print. PMID 41201562